CLINICAL TRIAL: NCT06171035
Title: Use of 3D Printing High-fidelity Airway and Craniofacial Manikin as an Education Tool to Improve Learning Efficiency of Teaching Noninvasive Positive Pressure Ventilation
Brief Title: Use of 3D Printing High-fidelity Craniofacial Manikin to Teach Noninvasive Positive Pressure Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH111188
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Satisfaction, Personal
Keywords: 3D printing; medical education model; high-fidelity simulation; respiratory care
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional model group (Active Comparator): Received a regular learning
  Interventions: Other: Traditional model education
- 3D-printed high-fidelity craniofacial manikin model presention group (Experimental): Received a regular learning plus 3D printing model
  Interventions: Other: 3D-printed high-fidelity craniofacial manikin model education

INTERVENTIONS:
Other: 3D-printed high-fidelity craniofacial manikin model education — Slide-based presention plus 3D printed model
  Arms: 3D-printed high-fidelity craniofacial manikin model presention group
Other: Traditional model education — Slide-based presention plus traditional model
  Arms: Traditional model group

SUMMARY:
The aim of this study is to enhance the learning efficiency and ability of problem-solving for student of Department of Respiratory Therapy with the innovative 3D printing high-fidelity manikin.

DETAILED DESCRIPTION:
Background :

Noninvasive positive pressure ventilation plays an important role in treatment of respiratory failure. Respiratory Therapists should be familiar with operating ventilator, choosing the adequate interface, and putting the interface on patients' face correctly. Simulation-based clinical training was limited because of lack of the high-fidelity manikins or simulators. To enhance the simulation-based clinical training, the investigators develop 3D printing models and applied into the medical school and hospital training.

Study Design :

The first part is a laboratory in-vitro experiment; the second part is a randomized controlled trial of medical education study.

Methods :

The 3D scanning and 3D printing technology will be using to create the high-fidelity manikin with an upper and lower airway tract. The 3D printing material will be choosing to be able to close real human organ especially considering the soft biological tissue. The present study will be divided into two parts. The first part is a laboratory in-vitro experiment, which aims to verified the function of the high-fidelity manikin; the second part is a medical education study.

Effect :

The investigators expect the use of 3D high-fidelity model in training students of Department of Respiratory Therapy will enhance the learning efficiency and ability of problem-solving.

The experience and outcome of the study will further extent to medical school and hospital training.

Key words:

3D printing; medical education model; high-fidelity simulation; respiratory care.

ELIGIBILITY:
Inclusion Criteria:

* Student of Fu Jen Catholic University

Exclusion Criteria:

* Refused to participate in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Examination score of pre-intervention | pre-intervention
  score of pre-intervention (maximun 100 and minimum 0), higher means a better outcome.
Examination score of post-intervention | immediately after the intervention
  score of post-intervention (maximun 100 and minimum 0), higher means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No